CLINICAL TRIAL: NCT05175586
Title: Physiotherapeutic Case Reports in Frozen Shoulder Pathology: Clinical Trial
Brief Title: Physiotherapeutic Case Studies in Frozen Shoulder Pathology
Acronym: CH-Case
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GEMA LEÓN BRAVO (Other)
Responsible Party: Sponsor-Investigator, GEMA LEÓN BRAVO, Principal Investigator, Clinica Gema Leon
Organization: Clinica Gema Leon (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ART-GLB-HOM-CONG; TFG-EFCH-2021 (Registry Identifier: TFG-EFCH-2021)
Record Dates: First submitted 2021-10-21; First posted 2022-01-04 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Articular; Rigid
Keywords: Stiff shoulder.; Neuromodulation.; Manual therapy.; Rotator cuff.; Physiotherapy.
MeSH Terms: conditions — Muscle Rigidity | interventions — Database Management Systems

STUDY DESIGN:
Intervention Model Description: 30 divided into two groups: Group 1 (n=15) percutaneous neuromodulation together with orthopaedic manual therapy (Maitland and Mulligan) Group 2 (n=15) orthopaedic manual therapy (Maitland and Mulligan).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): 15 patients in the experimental group of percutaneous neuromodulation together with orthopaedic manual therapy (Maitland and Mulligan)
  Interventions: Diagnostic Test: First data analysis; Procedure: Second data analysis; Other: database
- Group 2 (Active Comparator): 15 patients in the experimental group of orthopaedic manual therapy (Maitland and Mulligan).
  Interventions: Diagnostic Test: First data analysis; Procedure: Second data analysis; Other: database

INTERVENTIONS:
Diagnostic Test: First data analysis — A series of questions were asked to a number of patients with diagnoses related to primary idiopathic stiff shoulder and/or extrinsic stiff shoulder secondary to trauma or surgery. These patients are part of the physiotherapy clinic receiving the research. This questionnaire answers basic questions for the structure of the study such as age and sex, physical behaviour during the week, endurance, athletic disability, reason for attending the clinic, exploratory motor tests, etc. Subsequently, physiotherapeutic tests related to the pathology within the research were performed consisting of joint range, percentage of shoulder disability and pain scale.
Procedure: Second data analysis — Three treatment sessions of Percutaneous Neuromodulation (PNM) and Orthopaedic Manual Therapy (OMT) (Maitland and Mulligan) (group 1) and three treatment sessions of Orthopaedic Manual Therapy (OMT) (Maitland and Mulligan) (group 2) were performed at a rate of two sessions per month for three months. These therapies were compared with the clinical examination performed prior to each new session to verify changes in joint range, percentage of shoulder disability, strength and pain scale.
Other: database — Age and sex were expressed as mean ± standard deviation (SD). The rest of the variables were expressed as mean, absolute and relative frequency. The chi-square test was used to analyse the differences between the examinations in terms of the time taken and the treatments used in the two groups. A confidence level of 95% was established, considering a value of p<0.05 as statistically significant.

SUMMARY:
The stiff shoulder presents symptoms such as pain, loss of mobility and strength, being more common the idiopathic origin associated to the female gender. The definitive diagnosis presents complications due to the number of etiologies that can cause it. Epidemiologically, it presents from 2 to 5% of medical incapacities in the working population. Objective: To investigate the efficacy of percutaneous Neuromodulation together with Orthopedic Manual Therapy (Maitland and Mulligan) in comparison with Orthopedic Manual Therapy (Maitland and Mulligan) used in stiff shoulder.Design: Experimental clinical trial in 30 patients aged 21 to 76 years from a physiotherapy center divided into two groups: Group 1 (n=15) Percutaneous Neuromodulation + Orthopaedic Manual Therapy (Maitland and Mulligan) Group 2 (n=15) Orthopaedic Manual Therapy (Maitland and Mulligan).

DETAILED DESCRIPTION:
The stiff shoulder is a pathology characterized by a biomechanical restriction of the active and passive movement of the shoulder, showing clinical pictures of local inflammation with a notorious hyper vascularization that helps the clinical manifestations painful flexion, stiffness, limitation of external rotation, pain over the lower cervical area or near the insertion of the deltoid muscle and pain when supporting the affected limb with body weight.

Etiologically there are idiopathic and external factors that cause disorders such as osteoarthritis, chronic subacromial bursitis, or rotator cuff tendinopathy. Likewise, trauma is involved in a secondary way as well as diseases such as Parkinson's, diabetes, thyroid disorders among others. These clinical factors present two types of diagnosis: primary idiopathic stiff shoulder and extrinsic stiff shoulder secondary to trauma or surgery.

Among the physiotherapeutic treatments provided are joint mobilizations, therapeutic exercises, deep Cyriax massage, osteopathic techniques, cryotherapy (inflammatory phase), thermotherapy (chronic phase), electrotherapy for pain and ultrasound.

From the economic point of view, it presents from 2 to 5% of the medical incapacities in the working population, being this disease one of the first 20 sick leaves that reaches up to 12 months, generating high public hospital expenses and difficulties for the business area. Due to the above, many patients enter the operating room as a quick option to return to normality. However, this option does not seem to be the best for this disease, since the hypomobility of the movement increases gradually and chronically, caused by the fibrotic processes in the anterior face of the capsule, generating long-term inability for the external rotation of the joint.

The aim of this study is to investigate the efficacy of Percutaneous Neuromodulation together with Orthopaedic Manual Therapy (Maitland and Mulligan) compared to Orthopaedic Manual Therapy (Maitland and Mulligan) used in the stiff shoulder.

ELIGIBILITY:
Inclusion Criteria:

* Patients with difficulty in activities of daily living ABVD 35.
* Patients with positive results in some of the physical examination tests.
* Patients with a previous diagnosis by ultrasound imaging.
* Patients with surgical intervention after 3 months of age.

Exclusion Criteria:

* Patients with mental disorders or deficits.
* Patients with needle phobia (belonephobia).
* Patients with recent surgery before 3 months of age.
* Patients with previous dislocation of the affected shoulder.

Ages: 21 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
Pain scale (EVA) | 3 months
  The values of pain levels during the examination are reflected as follows:
  0= No pain 1-2= Little pain 3-4= Moderate pain 5-6= Severe pain 7-8= Very severe pain 9-10= Unbearable pain
Rigid shoulder type | 3 months
  Information on the type of stiff shoulder you have.
Daniels Scale | 3 months
  Muscle function values during the scan are reflected as follows, with 0 being a negative value and 5 a positive value:
  0= Muscle does not contract.
  1. Muscle contracts, but there is no movement.
  2. Muscle contracts and moves normally, but without resistance.
  3. Muscle contracts and resists to a good degree.
  4. Muscle contracts and resists to almost its full extent.
  5. The muscle contracts and resists at full amplitude.
Joint range | 3 months
  The values of joint range during the examination are reflected by means of the joint range scale which emphasizes specific degrees for elevation, external rotation and internal rotation.

SECONDARY OUTCOMES:
Number of participants in each physical therapy application | 3 months
  Three reviews were carried out corresponding to the three months of treatment. During these three months, participants received two sessions per week, for a total of 24 sessions:
  * Group 1 (n=15) received the percutaneous neuromodulation treatment together with orthopedic manual therapy (Maitland and Mulligan).
  * Group 2 (n=15) received orthopedic manual therapy treatment (Maitland and Mulligan) only.

CONTACTS AND LOCATIONS:
Overall Officials: Gema León Bravo, Physiotherap, Principal Investigator — Departamento de Enfermería, Farmacología y Fisioterapia, Universidad de Córdoba, Córdoba, España; Jaime Rando Anaya, Physiotherap, Study Chair — Universidad de Córdoba
Locations (1):
- Gema León Physiotherapy and Rehabilitation Clinic, Córdoba, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No
The request for the data will be studied and considered upon prior and justified request.

REFERENCES:
- [Background] Hiscock N, Bell S, Coghlan J. Pain, depression and the postoperative stiff shoulder. BMC Musculoskelet Disord. 2015 Dec 4;16:376. doi: 10.1186/s12891-015-0841-6. PMID 26637238
- [Background] Green HD, Jones A, Evans JP, Wood AR, Beaumont RN, Tyrrell J, Frayling TM, Smith C, Weedon MN. A genome-wide association study identifies 5 loci associated with frozen shoulder and implicates diabetes as a causal risk factor. PLoS Genet. 2021 Jun 10;17(6):e1009577. doi: 10.1371/journal.pgen.1009577. eCollection 2021 Jun. PMID 34111113
- [Background] Pandey V, Madi S. Clinical Guidelines in the Management of Frozen Shoulder: An Update! Indian J Orthop. 2021 Feb 1;55(2):299-309. doi: 10.1007/s43465-021-00351-3. eCollection 2021 Apr. PMID 33912325
- [Background] Challoumas D, Biddle M, McLean M, Millar NL. Comparison of Treatments for Frozen Shoulder: A Systematic Review and Meta-analysis. JAMA Netw Open. 2020 Dec 1;3(12):e2029581. doi: 10.1001/jamanetworkopen.2020.29581. PMID 33326025
- [Background] Akbar M, McLean M, Garcia-Melchor E, Crowe LA, McMillan P, Fazzi UG, Martin D, Arthur A, Reilly JH, McInnes IB, Millar NL. Fibroblast activation and inflammation in frozen shoulder. PLoS One. 2019 Apr 23;14(4):e0215301. doi: 10.1371/journal.pone.0215301. eCollection 2019. PMID 31013287
- [Background] Chan HBY, Pua PY, How CH. Physical therapy in the management of frozen shoulder. Singapore Med J. 2017 Dec;58(12):685-689. doi: 10.11622/smedj.2017107. PMID 29242941
- [Background] Ryan V, Brown H, Minns Lowe CJ, Lewis JS. The pathophysiology associated with primary (idiopathic) frozen shoulder: A systematic review. BMC Musculoskelet Disord. 2016 Aug 15;17(1):340. doi: 10.1186/s12891-016-1190-9. PMID 27527912
- [Background] Jeong, JY, Shim, SB, Hong, JH, Im, W., Lee, SM y Yoo, JC (2020). Efecto del hombro congelado preoperatorio sobre los resultados clínicos después de la reparación artroscópica del manguito rotador. Revista ortopédica de medicina deportiva , 8 (7), 2325967120934449. https://doi.org/10.1177/2325967120934449
- [Background] Cho, CH, Bae, KC y Kim, DH (2019). Estrategia de tratamiento para hombro congelado. Clínicas de cirugía ortopédica , 11 (3), 249-257. https://doi.org/10.4055/cios.2019.11.3.249
- [Background] Cui, J., Lu, W., He, Y., Jiang, L., Li, K., Zhu, W. y Wang, D. (2017). Biología molecular de la limitación inducida por el hombro congelado de los movimientos de la articulación del hombro. Revista de investigación en ciencias médicas: la revista oficial de la Universidad de Ciencias Médicas de Isfahan , 22 , 61. https://doi.org/10.4103/jrms.JRMS_1005_16
- [Background] Vastamäki, H., Ristolainen, L. y Vastamäki, M. (2016). El rango de movimiento del hombro congelado diabético se recupera al nivel contralateral. Revista de investigación médica internacional , 44 (6), 1191-1199. https://doi.org/10.1177/0300060516675112
- [Background] Uppal, HS, Evans, JP y Smith, C. (2015). Hombro congelado: una revisión sistemática de las opciones terapéuticas. Revista mundial de ortopedia , 6 (2), 263-268. https://doi.org/10.5312/wjo.v6.i2.263
- [Background] Park, EW, Cho, JH, Cho, CH, Sung, DH y Kim, DH (2021). Comparación de evaluaciones ecográficas de hombro entre polimialgia reumática y hombro congelado en pacientes con dolor de hombro bilateral: un estudio retrospectivo comparativo. Revista de medicina personalizada ,
- [Background] Dyer, BP, Burton, C., Rathod-Mistry, T., Blagojevic-Bucknall, M. y van der Windt, DA (2021). La diabetes como factor pronóstico en el hombro congelado: una revisión sistemática. Archivos de investigación en rehabilitación y traducción clínica , 3 (3), 100141. https://doi.org/10.1016/j.arrct.2021.100141
- [Background] Song, C., Song, C. y Li, C. (2021). Resultado de la manipulación bajo anestesia con o sin inyección de esteroides intraarticulares para el tratamiento del hombro congelado: un estudio de cohorte retrospectivo. Medicina , 100 (13), e23893. https://doi.org/10.1097/MD.0000000000023893